CLINICAL TRIAL: NCT05644665
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of Oral Ozanimod to Evaluate Efficacy and Long-term Safety in Chinese Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Brief Title: A Study to Evaluate Efficacy and Long-term Safety of Oral Ozanimod in Chinese Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM047-010
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Ozanimod (Experimental)
  Interventions: Drug: Ozanimod
- Arm B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Other Names: BMS-986374
  Arms: Arm A: Ozanimod
Drug: Placebo — Specified dose on specified days
  Arms: Arm B: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ozanimod compared with placebo in participants with ulcerative colitis (UC) in mainland China and Taiwan. The main study is composed of an induction period, maintenance period, safety follow-up, and participants meeting certain criteria will be given the opportunity to participate in an optional open label extension.

ELIGIBILITY:
Inclusion Criteria:

Main Study:

* Eligible participants must be Chinese.
* Participant has had moderately to severely active UC diagnosed at least 3 months prior to first investigational product administration.

Open-label Extension Period:

* Participants who have completed the Week 10 Visit and are non-responders at Week 10.
* Participants who have completed the Induction Period and entered the Maintenance Period experienced disease relapse during the Maintenance Period, or who have completed the Maintenance Period at Week 52.

Exclusion Criteria:

Main Study and Open-label Extension Period:

* Participant has severe extensive colitis, diagnosis of CD, indeterminate colitis, presence or history of a fistula consistent with CD, microscopic colitis, radiation colitis, or ischemic colitis.

Open-label Extension Period:

* Participant has clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, psychiatric, or other major systemic disease making implementation of the protocol or interpretation of the study difficult or that would put the participant at risk by continuing the study or that would have required a participant to discontinue treatment were observed during the Induction Period or Maintenance Period.
* Participant has clinically relevant cardiovascular conditions, including history or presence of recent myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, Class III/IV heart failure, sick sinus syndrome, or severe untreated sleep apnea were observed during the Induction Period or Maintenance Period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with clinical remission as measured by the 3-component Mayo Score | At week 10

SECONDARY OUTCOMES:
Proportion of participants with clinical remission as measured by the 3-component Mayo Score | At week 52
Proportion of participants with clinical response as measured by the 3-component Mayo Score | At week 10 and at week 52
Proportion of participants with endoscopic improvement | At week 10 and at week 52
Proportion of participants achieving histologic remission | At week 10 and at week 52
Proportion of participants with mucosal healing | At week 10 and at week 52
Proportion of participants in remission as measured by the 3-component Mayo Score while off corticosteroids for ≥ 12 weeks | At week 52
Proportion of participants with Treatment Emergent Adverse Events (TEAEs) | Up to 78 weeks
Proportion of participants with Serious Adverse Events (SAEs) | Up to 78 weeks
Proportion of participants with TEAEs leading to discontinuation of investigational product | Up to 78 weeks
Proportion of participants with TEAEs of special interest | Up to 78 weeks
Proportion of participants with clinical laboratory abnormalities | Up to 78 weeks
Proportion of participants with vital sign abnormalities | Up to 78 weeks
Proportion of participants with electrocardiogram (ECG) abnormalities | Up to 78 weeks
Proportion of participants with pulmonary function test abnormalities | Up to 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (51):
- China (43):
  - Local Institution - 0012, Hefei, Anhui
  - Local Institution - 0013, Wuhu, Anhui
  - Local Institution - 0052, Beijing, Beijing Municipality
  - Local Institution - 0050, Chongqing, Chongqing Municipality
  - Local Institution - 0011, Xiamen, Fujian
  - Local Institution - 0020, Guangzhou, Guangdong
  - Local Institution - 0036, Guangzhou, Guangdong
  - Local Institution - 0028, Guangzhou, Guangdong
  - Local Institution - 0019, Guangzhou, Guangdong
  - Local Institution - 0008, Guangzhou, Guangdong
  - Local Institution - 0004, Zhanjiang, Guangdong
  - Local Institution - 0051, Guilin, Guangxi
  - Local Institution - 0007, Shijiazhuang, Hebei
  - Local Institution - 0006, Shijiazhuang, Hebei
  - Local Institution - 0040, Wuhan, Hubei
  - Local Institution - 0037, Wuhan, Hubei
  - Local Institution - 0033, Wuhan, HUB
  - Local Institution - 0027, Changsha, Hunan
  - Local Institution - 0022, Changsha, Hunan
  - Local Institution - 0061, Changzhou, Jiangsu
  - Local Institution - 0046, Changzhou, Jiangsu
  - Local Institution - 0024, Nanjing, Jiangsu
  - Local Institution - 0045, Nanjing, Jiangsu
  - Local Institution - 0018, Suzhou, Jiangsu
  - Local Institution - 0009, Suzhou, Jiangsu
  - Local Institution - 0044, Wuxi, Jiangsu
  - Local Institution - 0042, Zhenjiang, Jiangsu
  - Local Institution - 0010, Shenyang, Liaoning
  - Local Institution - 0029, Xi'an, Shaanxi
  - Local Institution - 0026, Xi'an, Shaanxi
  - Local Institution - 0039, Jinan, Shandong
  - Local Institution - 0035, Shanghai, Shanghai Municipality
  - Local Institution - 0041, Shanghai, Shanghai Municipality
  - Local Institution - 0034, Shanghai, Shanghai Municipality
  - Local Institution - 0015, Taiyuan, Shanxi
  - Local Institution - 0032, Chengdu, Sichuan
  - Local Institution - 0025, Chengdu, Sichuan
  - Local Institution - 0031, Tianjin, Tianjin Municipality
  - Local Institution - 0047, Tianjin, Tianjin Municipality
  - Local Institution - 0049, Kunming, Yunnan
  - Local Institution - 0030, Hangzhou, Zhejiang
  - Local Institution - 0048, Fuzhou
  - Local Institution - 0053, Shanghai
- Taiwan (8):
  - Local Institution - 0054, Changhua County, Changhua
  - Local Institution - 0060, Taipei City, Taipei
  - Local Institution - 0058, New Taipei City
  - Local Institution - 0001, Taichung
  - Local Institution - 0059, Taichung
  - Local Institution - 0056, Taipei
  - Local Institution - 0057, Taipei
  - Local Institution - 0055, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com